CLINICAL TRIAL: NCT05043623
Title: Diagnosis of Respiratory Viruses in Children With Rhinoswab Junior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: Rhinomed Pty Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: HREC/77305/RCHM-2021
Record Dates: First submitted 2021-08-26; First posted 2021-09-14 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: SARS CoV 2 Infection; COVID-19
Keywords: Rhinoswab Junior
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: The study is organised sequentially into three phases due to research capacity
  Phase 1: The first 250 participants (5-18 years) will be randomly assigned to Arm 1 and Arm 2 for the clinician collected/supervised phase.
  Phase 2: 50 participants (5-18 years) will be allocated to Arm 3 for the self-collected Rhinoswab/saliva/combined nose+throat swab.
  Phase 3: 50 subsequent participants (1m - 5 years) will be allocated to Arm 4 for the self-collect throat+nose/saliva/RAT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm 1 - Clinician Collected/supervised Rhinoswab first, then CTDN swab (Experimental): Rhinoswab test administered and immediately followed by CTDN. Rhinoswab swab tested on respiratory panel vs CTDN swab tested on respiratory panel (standard of care).
  Interventions: Device: Rhinoswab Junior; Device: Combined nose and throat swab
- Arm 2 - Clinician Collected/supervised CTDN swab first, then Rhinoswab (Experimental): CTDN test administered and immediately followed by Rhinoswab. CTDN swab tested on respiratory panel (standard of care) vs Rhinoswab swab tested on respiratory panel.
  Interventions: Device: Rhinoswab Junior; Device: Combined nose and throat swab
- Arm 3 - Self-collected Rhinoswab, saliva swab, CTDN (Experimental): In children 5-18 years, the child/parent/guardian collects the three samples, in order of patient/parent preference. All samples will be tested on the SARS-CoV-2 laboratory panel (Allplex™ SARS-CoV-2 Assay - Seegene Inc)
  Interventions: Device: Rhinoswab Junior; Device: Combined nose and throat swab; Device: Saliva swab
- Arm 4 - Self-collected RAT, saliva, CTDN (Experimental): In children 1 month -5 years, the child/parent/guardian collects the three samples, in order of patient/parent preference. Saliva and CTDN samples will be tested on the SARS-CoV-2 laboratory panel (Allplex™ SARS-CoV-2 Assay - Seegene Inc), RAT test kit will be Abbott PanBio
  Interventions: Device: Combined nose and throat swab; Device: Saliva swab; Diagnostic Test: Abbott Panbio™ COVID-19 antigen self-test kit

INTERVENTIONS:
Device: Rhinoswab Junior — Rhinoswab Junior is a single use self-administered nasal swab intended to collect clinical specimens from the patient's nasal passages
  Arms: Arm 1 - Clinician Collected/supervised Rhinoswab first, then CTDN swab; Arm 2 - Clinician Collected/supervised CTDN swab first, then Rhinoswab; Arm 3 - Self-collected Rhinoswab, saliva swab, CTDN
Device: Combined nose and throat swab — Combined nose and throat swab (standard of care)
Device: Saliva swab — Saliva swab
  Arms: Arm 3 - Self-collected Rhinoswab, saliva swab, CTDN; Arm 4 - Self-collected RAT, saliva, CTDN
Diagnostic Test: Abbott Panbio™ COVID-19 antigen self-test kit — COVID-19 antigen self-test kit for the screening of active COVID-19 infection. It is a single-use, in vitro, visually read rapid immunoassay that uses a human nasal swab specimen for the qualitative detection of nucleocapsid protein SARS-CoV-2 antigen. It is intended to be used manually by untrained lay users (self testing) in a private setting.
  Arms: Arm 4 - Self-collected RAT, saliva, CTDN

SUMMARY:
A study to investigate Rhinoswab as an alternative method to combined throat and deep nasal (CTDN) swab for respiratory sample collection in children who present to the Royal Children's Hospital (RCH) for viral testing. Children and their parent/guardian will answer a short survey about their preferences. Laboratory staff will answer a short survey about handling the different samples.

DETAILED DESCRIPTION:
The microbiological test of choice for detection of respiratory viruses is a reverse transcription polymerase chain reaction (RT-PCR). The test is reported as "detected" or "not-detected" to the clinician. The Ct-value is a microbiological analysis that represents the number of amplification cycles required for a target gene to exceed a threshold level, to determine a negative or positive result and is interpreted to detect respiratory viruses. The Ct-value is used to measure viral load.

SARS-CoV-2, the virus that causes COVID-19, is a respiratory virus of specific interest. SARS-CoV-2 is detected in the upper respiratory tract. National guidelines for diagnosing COVID-19 in Australia require a combined throat and deep nasal swab (CTDN). No other testing options are routinely recommended in Australia. However, research and international guidelines recommend nasal swabs alone for SARS-CoV-2 detection. The Center for Disease Control and Prevention (USA) currently recommend the use of an anterior nasal swab alone as a method for detection of SARS-CoV-2. A recent systematic review suggested nasal swabs are a clinically acceptable alternative specimen collection methods. In addition to satisfactory diagnostic performance, nasal swabs are potentially less invasive, and can be self-collected.

Research at the Melbourne Children's Campus has identified that the CTDN or nasopharyngeal swab, are uncomfortable and distressing for children. The fear of the test is a barrier for presentation to a health service for a SARS-CoV-2 test. Parental and child reluctance to undergo testing may impact the public health response, through under-identification of pediatric cases.

The Rhinoswab is a TGA (Therapeutic Goods Administration) approved anterior nasal swab for children and adults. The design of the Rhinoswab allows for standardisation of the site of biological sampling, as compared with CTDN swabs which are operator dependent. It is designed to be more comfortable and to collect nasal secretions for PCR testing. The Rhinoswab Junior is a smaller paediatric version that has novelty features which add interest and distraction. The child can use the swab themselves, allowing autonomy and control. The capture and elution efficiency of the Rhinoswab has been shown to be comparable, if not slightly superior, to the capture and elution efficiency to the commercially available Copan eSwab by VIDRL (Victorian Infectious Diseases Reference Laboratory) and GNOMIX analyses.

The RCH has completed over 30,000 tests in children throughout the COVID-19 Pandemic from March 2020 to June 2021 at the Respiratory Infection Clinic and Emergency Department. The RCH nurses and doctors are well placed to trial the Rhinoswab due to extensive experience in testing children, and have developed related clinical practice guidelines.

This trial aims to determine the following in children 5-18 years of age:

* To determine the sensitivity and specificity of the Rhinoswab compared to the standard CTDN swab, in detecting viruses on the respiratory panel
* To determine whether Rhinoswab is non-inferior to the standard CTDN swab by comparing Ct values
* To determine the sensitivity and specificity of the throat swab alone and deep nasal swab alone, compared with the CTDN, in detecting respiratory viruses
* To investigate the comfort and preference of the Rhinoswab compared to the CTDN swab.
* To investigate the laboratory handling of the Rhinoswab compared to the CTDN swab.
* To determine the sensitivity and specificity of the Rhinoswab compared to CTDN swab, and saliva, in detecting respiratory viruses including SARS-CoV-2.

In children 1 month to 5 years:

• To investigate sensitivity and specificity of Rapid Antigen Test (RAT) compared to CTDN swab and saliva test in detected SARS-CoV-2

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic and requiring a COVID-19 test at RCH or confirmed/suspected COVID-19 at home.
* Aged between 1 month -18 years old.
* Parent/guardian present.
* Parents/self are able to provide consent.

Exclusion Criteria:

* < 1 month or >18 years old.
* Recent head or neck surgery
* Inability (e.g. non-English speaking and if no interpreter is available) or unwillingness to consent

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 339 (Actual)
Dates: Start 2021-08-26 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-08-28 (Actual)

PRIMARY OUTCOMES:
Sensitivity of Rhinoswab compared with CTDN for 13 viruses on standard respiratory panel (Clinician collected/supervised) | 5 minutes from administering test
  The results (detected/not detected) on all 13 viruses on the standard respiratory panel from both the Rhinoswab and the standard swabs will be obtained, and the sensitivity of the Rhinoswab compared to the CTDN determined. Sensitivity is calculated only in the participants who tested positive for the respective virus using the CTDN swab and is calculated as the proportion patients who tested positive on the Rhinoswab among those who tested positive on the CTDN swab. 95% confidence intervals will be calculated.
Specificity of Rhinoswab compared with CTDN for 13 viruses on standard respiratory panel (Clinician collected/supervised) | 5 minutes from administering test
  The results (detected/not detected) on all 13 viruses on the standard respiratory panel from both the Rhinoswab and the standard swabs will be obtained, and the specificity of the Rhinoswab compared to the CTDN determined. Specificity is calculated only in participants who tested negative for respiratory viruses and is calculated as the proportion patients who tested negative on Rhinoswab among those who tested negative on CTDN swab. 95% confidence intervals will be calculated.

SECONDARY OUTCOMES:
Ct-Value of respiratory viruses on Rhinoswab compared with Ct-value of respiratory viruses on CTDN (Clinician-Collected/Supervised) | 5 minutes from administering test
  Median Ct-Value of respiratory viruses on Rhinoswab compared with Ct-value of respiratory viruses on CTDN for each detection will be compared. The CT value for the undetected sample will be set at the maximum number of cycles performed in the laboratory (CT value maximum of 38.73). If the upper limit of the confidence interval is more than 3 Ct-value, the two swabs will be regarded as non-inferior.
Swab Preference Assessment (Clinician-Collected/Supervised ) | 5 minutes from administering test
  The preferability for the Rhinoswab, compared to the standard sample for respiratory virus testing is determined, using the Likert scale or picture-based chart for standardised responses. Descriptive analyses will be used to describe child/parent/research preferences.
  A) Child/parent/research nurse will be asked to rate comfort for each swab: Extremely Comfortable 1 to Extremely Uncomfortable 5 B) What is your preference for future testing between CTDN and Rhinoswab? C) Which swab was better CTDN vs Rhinoswab?
Median Ct-value of SARS-CoV-2 on Rhinoswab vs saliva vs CTDN (Self-collected) | 5 minutes from administering test
  Median Ct-Value of SARS-CoV-2 on Rhinoswab, saliva and CTDN will be compared. The CT value for the undetected sample will be set at the maximum number of cycles performed in the laboratory (CT value maximum of 38.73). If the upper limit of the 95% confidence interval for the median difference is less than 3 CT, the Rhinoswab will be regarded as non-inferior.
Sensitivity of Rhinoswab compared with CTDN for SARS-CoV-2 (Self-collected) | 5 minutes from administering test
  Sensitivity is calculated only in the participants who tested positive for SARS-CoV-2 using the CTDN swab and is calculated as the proportion patients who tested positive on the Rhinoswab among those who tested positive on the CTDN swab.
Specificity of Rhinoswab compared with CTDN for SARS-CoV-2 (Self-collected) | 5 minutes from administering test
  Specificity is calculated only in participants who tested negative for SARS-CoV-2and is calculated as the proportion patients who tested negative on Rhinoswab among those who tested negative on CTDN swab.
Comparison of RAT test (detected/not detected) to Ct-values for saliva and standard CTDN for SARS-CoV-2 only (Self-collected) | 15 minutes from administering test
  The SARS-CoV-2 results (detected/not detected) from the RAT test will be compared with Ct-values from saliva and standard CTDN swabs.
Sensitivity of RAT compared with saliva for SARS-CoV-2 only (Self-collected) | 15 minutes from administering test
  Sensitivity is calculated only in the participants who tested positive for SARS-CoV-2 using saliva and is calculated as the proportion patients who tested positive on RAT among those who tested positive on saliva.
Sensitivity of RAT compared to standard CTDN for SARS-CoV-2 only (Self-collected) | 15 minutes from administering test
  Sensitivity is calculated only in the participants who tested positive for SARS-CoV-2 using the CTDN swab and is calculated as the proportion patients who tested positive on RAT among those who tested positive on CTDN swab.
Laboratory handling assessment | 5 minutes for survey, to be completed up to 14 days post the last participant enrolled
  At the end of the study, the laboratory staff will be asked:
  A) Rate the handling experience of Rhinoswab vs CTDN using a Likert scale:
  Rhinoswab was easier to handle 1 to Rhinoswab was harder to handle 3 B) Was there a difference in processing the Rhinoswab versus the combined throat and deep nasal swab?: Rhinoswab was easier to process/There was no difference in processing/Rhinoswab was harder to process C) How did the Rhinoswab impact the workflow or lab efficiency compared to the standard combined throat and deep nasal swab?
  1 Very easy and no impact on workflow or lab efficiency to 5 Very difficult and many complications on workflow or lab efficiency D) What benefits or challenges, did you observe when working with Rhinoswab in the lab? (Freetext)

CONTACTS AND LOCATIONS:
Locations (1):
- Shidan Tosif, Parkville, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
Beginning 12 months following analysis and article publication, the following will be made available long-term for use by future researchers from a recognised research institution whose proposed use of the data has been ethically reviewed and approved by an independent committee and who accept MCRI's conditions for access:
  • Individual participant data that underlie the results reported in this article after de-identification (text, tables, figures and appendices).
Time Frame: Beginning 12 months following analysis and article publication

REFERENCES:
- [Derived] Tosif S, Lee LY, Nguyen J, Overmars I, Selman C, Grobler AC, McMinn A, Waller G, McNab S, Jarvis T, Steer A, Babl FE, Daley A, Crawford NW. A novel anterior nasal swab to detect respiratory viruses: a prospective study of diagnostic accuracy. BMC Pediatr. 2023 Apr 28;23(1):201. doi: 10.1186/s12887-023-03976-5. PMID 37106344
- [Derived] Tosif S, Lee LY, Nguyen J, McMinn A, Selman C, Grobler AC, Daley A, Crawford NW. Stick with the nose...Saliva rapid antigen testing is not a viable method for testing children under 5 years old. J Paediatr Child Health. 2023 Feb;59(2):258-263. doi: 10.1111/jpc.16277. Epub 2022 Nov 18. PMID 36401338